CLINICAL TRIAL: NCT02137031
Title: Continuous Glucose Monitoring and HbA1c in Children for Longterm Diabetes Management
Brief Title: Continuous Glucose Monitoring and Metabolic Control in Children With Type 1 Diabetes
Acronym: CHILD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Krystie Robinson-Vincent, PhD Candidate, University of Toronto
Purpose: Treatment
Other Study IDs: 27225
Record Dates: First submitted 2014-05-07; First posted 2014-05-13 (Estimated); Last update posted 2014-05-13 (Estimated); Status verified 2014-05

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Mini Link REAL-Time Transmitter (Experimental)
  Interventions: Device: Mini Link REAL-Time Transmitter

INTERVENTIONS:
Device: Mini Link REAL-Time Transmitter — Children used the Mini Link REAL-Time Transmitter to measure glucose continuously for a minimum of three days per week for three months.

SUMMARY:
The primary purpose of this pilot randomized controlled trial is to provide preliminary indicators of the effects of continuous subcutaneous insulin infusion with continuous glucose monitoring compared to self-monitoring of blood glucose alone on: (1) metabolic control and (2) fear of hypoglycemia. Additional objectives will be: (1) to provide an estimate of recruitment rates, (2) to assess compliance with allocated treatment, and (3) to determine participants' satisfaction with allocated treatment.

With increased and immediate information related to current and future (trend) glucose information provided by the continuous glucose monitor, children can then act upon this knowledge to prevent hypo- or hyperglycemia, thus, experiencing a reduction in glucose variability, leading to an improvement in metabolic control as shown by a reduction in HbA1c levels.

Research on the effectiveness of continuous glucose monitoring on metabolic control in children with T1D using continuous subcutaneous insulin infusion has been limited. Therefore, a pilot clinical trial will be designed to provide preliminary indicators of the feasibility and acceptability of continuous glucose monitoring on metabolic control and address the following objectives.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6-18 years
* T1D for greater than one year;
* Willing to perform at least three self-monitoring blood glucose tests per day;
* Has been using continuous subcutaneous insulin infusion for more than one month
* English speaking

Exclusion Criteria:

* Presence of celiac disease (can cause malabsorption of nutrients affecting metabolic control)
* Use of corticosteroids that have systemic effects and affect glucose levels
* Currently using continuous glucose monitoring
* Cognitively unable to self-manage, based on parent's and/or care provider's opinion

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2012-09; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
HbA1c | 3 months
  Metabolic control as measured by standard HbA1c

SECONDARY OUTCOMES:
Fear of Hypoglycemia | 3 months
  Fear of Hypoglycemia as measured by Children's Hypoglycemia Index
Frequency of Hypoglycemia | 3 months
  The number of hypoglycemic episodes experienced per person over three months
Frequency of Hyperglycemia | 3 months
  Number of hyperglycemic episodes per person over the course of 3 months
Frequency of Diabetic Ketoacidosis | 3 months
  Frequency of Diabetic Ketoacidosis episodes per person over the course of 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Krystie A Robinson-Vincent, PhD c, Principal Investigator — University of Toronto
Locations (2):
- Canada (2):
  - Royal Victoria Hospital, Barrie, Ontario
  - Charles H. Best Centre, Whitby, Ontario